CLINICAL TRIAL: NCT02179424
Title: Assessing the Corporate Environment in Promoting Tobacco Control and Evaluation of a Smoking Cessation Programme in Workplaces in Hong Kong
Brief Title: Promoting Tobacco Control and Smoking Cessation in Workplaces [Phase I]
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Lok Sin Tong Benevolent Society, Kowloon (Other)
Responsible Party: Principal Investigator, Professor Lam Tai-Hing, Chair Professor and Director, School of Public Health, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LSTWPLACE
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Results first posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-10

CONDITIONS: Smoking
Keywords: smoking cessation interventions
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Health talk + Workshop + Booklet + SMS (Experimental): Health talk + workshop (Motivational intervention) + booklet + Short Message Service (SMS)
  Interventions: Behavioral: Workshop
- Face-to-face counseling + Booklet + SMS (Experimental): Face to Face counseling (Motivational intervention) + Booklet + SMS
  Interventions: Behavioral: Face-to-face counseling; Behavioral: Booklet; Behavioral: SMS
- Phone counseling + Health talk + Booklet + SMS (Experimental): Phone counseling (Motivational intervention) + Health talk + booklet + SMS
  Interventions: Behavioral: Phone counseling; Behavioral: Health talk; Behavioral: Booklet; Behavioral: SMS
- Phone counseling + Booklet + SMS (Experimental): Phone counseling (Motivational intervention) + booklet + SMS
  Interventions: Behavioral: Phone counseling; Behavioral: Booklet; Behavioral: SMS

INTERVENTIONS:
Behavioral: Workshop — Intensive psychological intervention included motivation of quitting enhancement, stress management and smoking triggers, craving and relapse are used to provide smoking cessation intervention
  Arms: Health talk + Workshop + Booklet + SMS
Behavioral: Face-to-face counseling — Use motivational interview strategies through face-to-face counseling to provide smoking cessation intervention
  Arms: Face-to-face counseling + Booklet + SMS
Behavioral: Phone counseling — Use motivational interview strategies through phone counseling to provide smoking cessation intervention.
  Arms: Phone counseling + Booklet + SMS; Phone counseling + Health talk + Booklet + SMS
Behavioral: Health talk — Health talk provided information about hazards of tobacco (active smoking, second- and third-hand smoke), benefits of quitting smoking and methods to quit smoking.
  Arms: Phone counseling + Health talk + Booklet + SMS
Behavioral: Booklet — A 26-page booklet included information about smoking and diseases, benefits of quitting smoking, methods to quit smoking, how to handle withdrawal symptoms, stress management, declaration of quitting smoking, decisional balance of smoking or quitting.
  Arms: Face-to-face counseling + Booklet + SMS; Phone counseling + Booklet + SMS; Phone counseling + Health talk + Booklet + SMS
Behavioral: SMS — Fifteen SMS were sent to subjects included welcome messages, risk of smoking, correction of myths about smoking or quitting, quitting tips, benefits of quitting, encouragement of quitting
  Arms: Face-to-face counseling + Booklet + SMS; Phone counseling + Booklet + SMS; Phone counseling + Health talk + Booklet + SMS

SUMMARY:
Previous research shows a significant proportion of smokers work in full-time employment. Given that the majority of smokers do not aware of the smoking cessation services available in Hong Kong, implementing smoking cessation policy in the workplaces may assist a considerable number of smokers to stop or reduce smoking.

This study aims to:

1. examine the employers' knowledge, attitudes and practices in promoting smoking cessation in workplace.
2. test the effectiveness of a brief and an intensive smoking cessation interventions to help workers stop smoking

In Phase I of this study, a large scale cross-sectional survey will be conducted to 3000 corporate companies in Hong Kong. The questionnaire will examine the employers' knowledge, attitudes and practices in promoting smoking cessation in the workplaces.

In Phase II, a longitudinal study will be conducted to evaluate the effectiveness of a smoking cessation intervention offered by the Department of Psychology, the University of Hong Kong. Smokers from the participating companies will be interviewed before the intervention at baseline, immediately after the intervention, and at 1-, 4-, 12-, 26- and 52-week post-intervention follow-ups.

The follow-up assessments will consist of a biochemical validation for the self-reported quitters who report quitting in the past 7 days via exhaled carbon monoxide and saliva cotinine concentration tests. Participants' smoking behaviour, knowledge on smoking and satisfaction of the smoking cessation services will also be evaluated.

It is hypothesized that the smoking cessation intervention helps workers stop smoking. Employers' knowledge and attitudes are positively associated with the practices in promoting smoking cessation in workplace.

Process evaluation: Qualitative interviews, including in-depth interviews and/or focus group will be conducted after 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 or above
* Cantonese speaker and able to read in Chinese characters
* Smoke at least one cigarette per day
* Stay at Hong Kong during the intervention and follow-up periods (12 months)

Exclusion Criteria:

* Smokers who are psychologically or physically unable to communicate
* Smokers who are currently following other smoking cessation programme(s)
* Smokers with diagnosed psychiatric illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Actual)
Dates: Start 2012-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tai Hing Lam, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- 2/F, 61 Lung Kong Rd, Kowloon City, Lok Sin Tong Benevolent Society, Hong Kong, China

REFERENCES:
- [Derived] Wang MP, Li WHC, Suen YN, Cheung KC, Lau OS, Lam TH, Chan SSC. Association between employer's knowledge and attitude towards smoking cessation and voluntary promotion in workplace: a survey study. Tob Induc Dis. 2017 Nov 14;15:44. doi: 10.1186/s12971-017-0149-4. eCollection 2017. PMID 29162997
- [Derived] Wang MP, Suen YN, Li WHC, Lau OS, Lam TH, Chan SSC. Proactive outreach smoking cessation program for Chinese employees in China. Arch Environ Occup Health. 2018 Mar 4;73(2):67-78. doi: 10.1080/19338244.2017.1308309. Epub 2017 Apr 21. PMID 28350250

RESULTS

PARTICIPANT FLOW:
Groups:
- Health Talk + Workshop + Booklet + SMS: Health talk + workshop (Motivational intervention) + booklet + Short Message Service (SMS)
  Motivational intervention: Use motivational interview strategies to provide smoking cessation intervention
- Face-to-face Counseling + Booklet + SMS: Face to Face counseling (Motivational intervention) + Booklet + SMS
  Motivational intervention: Use motivational interview strategies to provide smoking cessation intervention
- Phone Counseling + Health Talk + Booklet + SMS: Phone counseling (Motivational intervention) + Health talk + booklet + SMS
  Motivational intervention: Use motivational interview strategies to provide smoking cessation intervention
- Phone Counseling + Booklet + SMS: Phone counseling (Motivational intervention) + booklet + SMS
  Motivational intervention: Use motivational interview strategies to provide smoking cessation intervention
Period: Overall Study
Arm/Group | Health Talk + Workshop + Booklet + SMS | Face-to-face Counseling + Booklet + SMS | Phone Counseling + Health Talk + Booklet + SMS | Phone Counseling + Booklet + SMS
Started | 76 | 11 | 516 | 39
Completed | 76 | 11 | 516 | 39
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: Health talk + workshop (Motivational intervention) + booklet + Short Message Service (SMS)
  Motivational intervention: Use motivational interview strategies to provide smoking cessation intervention
- Group B: Face to Face counseling (Motivational intervention) + Booklet + SMS
  Motivational intervention: Use motivational interview strategies to provide smoking cessation intervention
- Group C: Phone counseling (Motivational intervention) + Health talk + booklet + SMS
  Motivational intervention: Use motivational interview strategies to provide smoking cessation intervention
- Group D: Phone counseling (Motivational intervention) + booklet + SMS
  Motivational intervention: Use motivational interview strategies to provide smoking cessation intervention
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Total
Number analyzed (Participants) | 76 | 11 | 516 | 39 | 642
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.8 (28.5) | 51.1 (19.3) | 81.5 (28.0) | 60.0 (26.6) | 78.9 (28.6)
Gender [Count of Participants; unit: Participants]
  Female | 9 | 1 | 89 | 4 | 103
  Male | 67 | 10 | 427 | 35 | 539
Region of Enrollment [Number; unit: participants]
  China | 76 | 11 | 516 | 39 | 642

OUTCOME MEASURES:

1. Primary Outcome: Employers' KAP
Description: A questionnaire aimed to examine the employers'/ managerial staff's knowledge, attitudes and practices in promoting smoking cessation in the workplace.
  The questionnaires consist of three parts:
  1. Employers's knowledge was assessed by measuring the average number of correct answers on questions about smoking and quitting (Scale 1-7).
  2. Employers' attitude was assessed by measuring the average number agreeing items about their willingness to support employees to quit which included implementation of measures to show support for smoking cessation in the workplace or participation in smoking cessation programme (Scale 1-17).
  3. Employers' practice was assessed by the level of smoking ban in the workplace as reported by the employer. (Scale 1-4; 1: not prohibited, 2: prohibited by not strictly, 3: Strictly prohibited and 4: absolutely strictly prohibited).
Time Frame: Before the health talk
Population: In Phase 1, questionnaires were sent out to 580 companies and 292 of the company employers returned the complete questionnaire. These 292 employers were not participating in the Phase 2 of this study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Employers' KAP: Employers' knowledge on smoking and quitting
Arm/Group | Employers' KAP
Number analyzed (Participants) | 292
units on a scale
  Employers' knowledge on smoking and quitting | 3.08 (3.24)
  Employers' attitude on assisting employees to quit | 6.06 (4.16)
  Employers' practice on smokefree workplace policy | 3.40 (0.76)

2. Primary Outcome: Smoking Quit Rate
Description: smoking quit rate was defined as the self-reported 7-day point prevalence abstinence
Time Frame: 6 month follow-up and 12 month follow-up
Population: In Phase 2, a sample of 642 employees enrolled in the study and chose 1 among the 4 conditions for smoking cessation.
Measure: Number; unit: participants
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 76 | 11 | 516 | 39
participants
  6-month Follow up | 26 | 3 | 155 | 15
  12-month Follow up | 29 | 4 | 164 | 14

3. Secondary Outcome: Smoking Reduction
Description: Reduced at least 50% of cigarette consumption
Time Frame: 6 month follow-up and 12 month follow-up
Measure: Number; unit: participants
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 76 | 11 | 516 | 39
participants
  6-month follow up | 16 | 5 | 70 | 5
  12-month follow up | 15 | 1 | 66 | 4

ADVERSE EVENTS:
Arm/Group | Group A | Group B | Group C | Group D
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/11 | 0/516 | 0/39
Other Adverse Events (participants affected / at risk) | 0/76 | 0/11 | 0/516 | 0/39

LIMITATIONS AND CAVEATS:
The study did not randomize subjects to the intervention groups and had no control group. The 4 groups could not be assumed to be comparable. The sample size of each group varied greatly, which undermined the predictive power of the interventions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No